CLINICAL TRIAL: NCT05325229
Title: A Single-arm, Multicenter, Phase II Clinical Study of Docetaxel for Injection (Albumin-bound) in Combination With Bevacizumab in Patients With Platinum-Resistant Recurrent Ovarian Cancer
Brief Title: A Study of Docetaxel for Injection (Albumin-bound) in Combination With Bevacizumab in Patients With Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB1801-005
Record Dates: First submitted 2022-03-24; First posted 2022-04-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-03

CONDITIONS: Platinum-resistant Recurrent Ovarian Cancer
MeSH Terms: interventions — Docetaxel; Injections; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Docetaxel combined with Bevacizumab (Experimental): Docetaxel for Injection (Albumin-bound) will be administrated once every 3 weeks at a dose of 75 mg/m^2 or 100 mg/m^2; Bevacizumab will be administrated once every 3 weeks at a dose of 15mg/kg.
  Interventions: Drug: Docetaxel for injection (Albumin-bound); Drug: Bevacizumab

INTERVENTIONS:
Drug: Docetaxel for injection (Albumin-bound) — Docetaxel for injection (Albumin-bound), by intravenous infusion，75 mg/m^2 or 100 mg/m^2 once every 3 weeks.
Drug: Bevacizumab — Bevacizumab, by intravenous infusion, 15 mg/kg once every 3 weeks.

SUMMARY:
This trial is a single-arm, multicenter clinical study to evaluate the efficacy and safety of Docetaxel for Injection (Albumin-bound) combined with Bevacizumab and the pharmacokinetic characteristics of Docetaxel in patients with platinum-resistant recurrent ovarian cancer.

DETAILED DESCRIPTION:
This study will be conducted in two stages (dose escalation trial and phase II trial). Dose escalation trial: To explore the safety and tolerability of Docetaxel for Injection (Albumin-bound) (75 mg/m^2 and 100 mg/m^2) combined with Bevacizumab 15 mg/kg. Dose escalation will be started at low dose and proceed in turn.

Phase II trial: According to the recommended phase II dose (RP2D) determined in the dose escalation trial, a phase II study of Docetaxel for Injection (Albumin-bound) combined with Bevacizumab will be conducted to observe the efficacy of the combination regimen, with overall response rate (ORR) as the primary study endpoint. Simon's optimal 2-stage design will be adopted for phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18, ≤78 years (subject to the date when the informed consent form is signed) and voluntarily signed the informed consent form.
2. Histologically or cytologically confirmed diagnosis of epithelial ovarian, fallopian tube, or primary peritoneal cancer.
3. Patients who responded to their last line of platinum treatment, and the disease recurred or progressed between 28 days to 6 months (184 calendar days) after the last platinum therapy (platinum-resistant disease), with no more than two lines of non-platinum therapy.
4. At least one measurable lesion according to RECIST v1.1.
5. Patients with Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
6. Patients with estimated survival time of ≥ 3 months.
7. Main organ function meets the following criteria within 7 days before treatment (no medical supportive treatments such as blood component transfusion, human granulocyte colony-stimulating factor (G-CSF), thrombopoietin (TPO), interleukin-11, and erythropoietin (EPO) within 2 weeks before administration of the investigational drug):

   Absolute neutrophil count ≥1.5×10^9/L; Platelets ≥100×10^9/L; Hemoglobin ≥90 g/L or ≥5.6 mmol/L; Serum creatinine ≤ 1.5×ULN or creatinine clearance rate ≥ 40 mL/min; Liver function: total bilirubin≤ 1.0 × ULN, ≤ 1.5 × ULN for patients with liver metastasis; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 × ULN, ≤ 2.5 × ULN for patients with liver metastasis.

   Activated Partial Thromboplastin Time (APTT) ≤ 1.5×ULN, International Normalized Ratio (INR) ≤ 1.5×ULN.
8. The patient must agree to take adequate contraception from signing of ICF through 6 months after last dose, women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to the first dose of the investigational drug.

Exclusion Criteria:

1. Patients who have received anti-angiogenic therapy (including but not limited to bevacizumab, apatinib, anlotinib, etc.) within 18 weeks before the first use of the investigational drug.
2. The progression-free interval of previous docetaxel treatment was less than 6 months.
3. Patients whose disease progressed during platinum therapy (from the first dose to 28 days after the last dose).
4. Mucinous ovarian cancer or less malignant ovarian tumors (such as low-grade serous ovarian cancer).
5. Symptomatic central nervous system (CNS) metastases or cancerous meningitis (Patients may participate in this study if they have completed radiotherapy or surgery for CNS metastases prior to screening, and the patient's nervous system has been stable for ≥4 weeks after radiotherapy or post-surgery (i.e., no new neurological deficits due to brain metastases, no new lesions on CNS imaging, and no treatment is required at screening)).
6. History of other malignant tumors within 5 years before the first dose of the investigational drug, except for the following: curable cancer such as basal cell or squamous cell skin cancer, superficial bladder cancer, prostate cancer, cervical cancer or breast cancer in situ that had been cured.
7. Patients with a history of thromboembolism, cerebral infarction, hemorrhagic disease or bleeding tendency within 6 months before the first dose of the investigational drug.
8. History of intestinal obstruction, gastrointestinal perforation, abdominal fistula or abdominal abscess within 6 months before the first dose of the investigational drug.
9. Abdominal or pelvic radiotherapy within 5 years before the first dose of the investigational drug.
10. Urine protein >2+, or urine protein is 2+ with 24-hour urine protein quantitative >1g at screening.
11. Patients who are known to be allergic to the investigational drug or its main excipients.
12. Patients with an uncontrollable third space effusion (e.g. pleural effusion, ascites, or pericardial effusion), who, in the judgment of the investigator, are not suitable for the study.
13. Patients with a history of severe cardiovascular disease, including but not limited to:

    1. Severe heart rhythm or conduction abnormalities, including but not limited to ventricular arrhythmia requiring clinical intervention and third degree atrioventricular block within 6 months before the first dose of the investigational drug;
    2. History of myocardial infarction, angina pectoris, angioplasty and coronary artery bypass surgery within 6 months before the first dose of the investigational drug;
    3. Heart failure with New York Heart Association (NYHA) Classification of Class III and above;
    4. Poorly controlled hypertension (Systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 95 mmHg at screening period despite optimal therapy);
    5. Patients with prolonged QT/QTc interval (QTcF > 480 ms, Fridericia's formula: QTcF = QT/RR^0.33, RR = 60/heart rate) during the screening period;
    6. Left ventricular ejection fraction (LVEF) <50% during the screening period.
14. HCV antibody (+) is positive during the screening period (HCV RNA negative can be included, anti-HCV treatment other than interferon is allowed), active hepatitis B disease (HBV DNA ≤2000 IU/mL can be included, anti-HBV treatment other than interferon is allowed), HIV positive, or with acquired immunodeficiency syndrome (AIDS).
15. Patients who have undergone major organ surgery within 4 weeks before the first dose of the investigational drug, or who need to undergo elective surgery during the study.
16. Adverse reactions from the previous anti-tumor treatment have not yet recovered to ≤ level 1 based on CTCAE 5.0 (except for the toxicity without safety risk judged by the investigator, such as Grade 2 neuropathy, alopecia).
17. Patients who have received anti-tumor treatments such as chemotherapy, targeted therapy, immunotherapy and other clinical study drugs within 4 weeks before the first dose of the investigational drug, and other conditions are as follows: Local palliative radiotherapy within 2 weeks before the first dose of the investigational drug; oral fluoropyrimidines, small molecule targeted drugs, etc. within 2 weeks before the first dose of the investigational drug or within known 5 half-lives of the drug (whichever is longer); Traditional Chinese medicines with anti-tumor indications within 2 weeks before the first dose of the investigational drug.
18. Patients who have used potent inhibitors or inducers of CYP3A4 within 2 weeks before the first dose of the investigational drug.
19. Patients who have received a live attenuated vaccine within 4 weeks before the first use of the investigational drug.
20. Patients who have taken aspirin (>325mg/day) or other non-steroidal anti-inflammatory drugs that may affect platelet function within 10 days before the first use of the investigational drug.
21. Nursing women.
22. Patients with active infection requiring intravenous antibiotic therapy (at the discretion of the investigator).
23. Patients with a history of alcohol or drug dependence.
24. Other situations that the investigator considers not suitable for participating in the clinical study, including but not limited to: the patient is complicated by severe or uncontrolled medical conditions, which interfere with the interpretation of study results and affect the study compliance.

Ages: 18 Years to 78 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 94 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Dose escalation trial: Incidence of adverse event(AE) | Up to approximately 2 years
Phase II trial: Overall response rate (ORR) by Independent Review Committee(IRC) | Up to approximately 2 years
Dose escalation trial: Serious adverse event(SAE ) | Up to approximately 2 years
Dose escalation trial: Dose limiting toxicity(DLT). | Up to approximately 2 years

SECONDARY OUTCOMES:
Dose escalation trial and Phase II trial: Plasma concentration of docetaxel (free and total | Up to approximately 3 months
Phase II trial: ORR by investigator | Up to approximately 2 years
Phase II trial: Disease control rate (DCR) | Up to approximately 2 years
Phase II trial: Duration of Response (DOR) | Up to approximately 2 years
Phase II trial: Progression-Free-Survival (PFS) | Up to approximately 2 years
Phase II trial: Overall survival (OS) | Up to approximately 2 years
Phase II trial: CA125 response rate | Up to approximately 2 years
  Proportion of patients with a minimum 50% reduction in CA125 serum levels lasting for 28 days relative to baseline CA-125 serum levels, for patients whose baseline CA-125 serum levels ≥2×ULN.
Phase II trial: Incidence of AE | Up to approximately 2 years
Phase II trial: abnormal vital signs | Up to approximately 2 years
Phase II trial: abnormal physical examination | Up to approximately 2 years
Phase II trial: abnormal electrocardiogram | Up to approximately 2 years
Phase II trial: abnormal laboratory tests | Up to approximately 2 years
Phase II trial: Eastern Cooperative Oncology Group（ECOG） scores | Up to approximately 2 years
  There are 6 values (0, 1,2,3,4,5) in the ECOG score system. A higher score means a worse outcome, for example, 0 means normal, 5 means death.

CONTACTS AND LOCATIONS:
Overall Officials: Xuekun Yao, Study Director — CSPC ZhongQi Pharmaceutical Technology Co., Ltd.
Locations (1):
- Tongji Hospital,Tongji Medical College of HUST, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided